CLINICAL TRIAL: NCT07188727
Title: Refining Clinical Practice in Ulcerative Colitis: The Prognostic Value of Histologic Remission - A Monocentric Retrospective Study
Brief Title: Comparative Outcomes of Ulcerative Colitis Patients With Mayo Endoscopic Score 1 and Histologic Activity Versus Mayo Endoscopic Score 2
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Ferdinando D'amico, MD, PhD, IRCCS San Raffaele
Other Study IDs: MES1VSMES2
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Ulcerative Colitis; Histology; Mayo Endoscopic Score; Outcomes
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mayo Endoscopic Score 1: Patients with ulcerative colitis who initiated advanced therapy and had mild endoscopic activity at baseline (Mayo Endoscopic Subscore 1). Histologic findings were recorded, and long-term outcomes such as surgery and hospitalization were assessed.
- Mayo Endoscopic Score 2: Patients with ulcerative colitis who initiated advanced therapy and had moderate endoscopic activity at baseline (Mayo Endoscopic Subscore 2). Long-term outcomes, including surgery and hospitalization, were evaluated for comparison with the MES1 group.

SUMMARY:
This retrospective study examines patients with ulcerative colitis who initiated advanced therapy for their disease. In clinical practice, patients with only mild inflammation on endoscopy (Mayo Endoscopic Subscore 1, or MES1) often do not undergo treatment optimization or therapy change. We stratified these patients based on histologic findings from biopsy samples and compared them with patients who had greater endoscopic activity (MES2). We evaluated long-term outcomes, including surgery and hospitalization, to determine whether current management strategies for patients with mild endoscopic disease should be reconsidered.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of UC (by routine clinical, radiographic, endoscopic and pathologic criteria);
* Patients starting a new advanced treatment for UC (either biologic agents or small molecules);
* Patients with endoscopic MES of 1 or 2 at the endoscopic reassessment (conducted after 12 ± 3 months following the initiation of advanced therapy)

Exclusion Criteria:

* Patients with unclassified colitis or Crohn's disease;
* Previous colonic surgery (eg. Pouch);
* Patients for whom biopsies were not obtained at the time of endoscopic reassessment (conducted after 12 months following the initiation of advanced therapy);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with ulcerative colitis who initiated advanced therapy between 2019 and 2025. Patients were stratified according to baseline Mayo Endoscopic Subscore (MES1 or MES2) and had available histologic assessment from endoscopic biopsies.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Composite Outcome | From enrollment to end of follow-up at 36 months
  The composite outcome includes any of the following events: escalation of medical therapy, hospitalization related to ulcerative colitis, or surgery related to ulcerative colitis

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, MI, Italy